CLINICAL TRIAL: NCT03606785
Title: Evaluation of the Efficacy and Safety of Single Dose Tranexamic Acid in Reducing Blood Loss During Colorectal Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201617010.2P
Record Dates: First submitted 2018-07-14; First posted 2018-07-31 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Surgery
Keywords: colorectal,blood, transfusion,haemorrhage,tranexamic acid.
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid group (Active Comparator)
  Interventions: Drug: Tranexamic Acid Injection
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo injection

INTERVENTIONS:
Drug: Tranexamic Acid Injection — The TA group will receive an intravenous bolus of (10 mg/kg) in 100 ml of normal saline over 20 minutes after induction of anesthesia and before surgical incision
  Arms: tranexamic acid group
Drug: placebo injection — patients will receive a placebo of 100 mL 0.9% normal saline
  Arms: placebo group

SUMMARY:
A total of 46 patients scheduled for explorative laparotomy with the aim of radical debulking surgery for colorectal cancer will be randomized into two equal groups one will receive tranexamic acid and one placebo.

The TA group will receive an intravenous bolus of (10 mg/kg) in 100 ml of normal saline over 20 minutes after induction of anesthesia and before surgical incision. In the control group, patients will receive a placebo of 100 mL 0.9% normal saline. The primary endpoint is reduction in blood loss, while the secondary endpoint was the number of patients needing transfusion and occurrence of postoperative thrombotic complications (myocardial infarction, stroke, pulmonary embolism, renal failure, or bowel infarction) within 30 days after surgery.

ELIGIBILITY:
Inclusion criteria

* ASA 1 and ASA 2 patients scheduled for colorectal cancer surgery.
* Age above 18 years & less than 65 years.

Exclusion criteria:

* Thrombophilia or any bleeding disorder.
* Previous or active thromboembolic disease.
* Family history of thromboembolism.
* Known Allergy to TA.
* Liver dysfunction.
* Preexisting renal dysfunction (serum creatinine >1.2 mg/dL).
* Coronary stent insertion within a year prior to operation.
* Cardiovascular problem (e.g., myocardial infarction, atrial fibrillation, angina, heart failure),
* Lifelong warfarin therapy for thromboembolism prophylaxis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
reduction in blood loss | 1 month
  Blood loss will be calculated (volume estimated as the blood remaining in sponges and drapes and the volume in suction bottles during surgery).The amount of drained blood will be measured in 1st 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- NCI, Cairo university, Cairo, Egypt